CLINICAL TRIAL: NCT00004164
Title: A Phase II Trial of Docetaxel, Cisplatin, 5-FU, and Leucovorin for Carcinoma of the Nasopharnyx
Brief Title: Combination Chemotherapy in Treating Patients With Stage IIB, Stage III, or Stage IV Cancer of the Nasopharynx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067408; DFCI-99132; RP-DFCI-99132; NCI-G99-1631
Record Dates: First submitted 1999-12-10; First posted 2004-07-19 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2000-09

CONDITIONS: Head and Neck Cancer
Keywords: stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms | interventions — Filgrastim; Cisplatin; Docetaxel; Fluorouracil; Leucovorin; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Drug: leucovorin calcium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have stage IIB, stage III, or stage IV cancer of the nasopharynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and overall response rate to docetaxel, cisplatin, fluorouracil, and leucovorin calcium in patients with potentially curable nasopharyngeal cancer. II. Assess the tolerability of this regimen in these patients.

OUTLINE: Patients receive docetaxel IV over 1 hour followed 1 hour later by cisplatin IV over 4 hours and fluorouracil IV and leucovorin calcium IV over 96 hours. Filgrastim (G-CSF) is administered subcutaneously beginning on day 5 and continuing until blood counts recover or day 10. Treatment repeats every 3 weeks for up to 3 courses. Within 2 weeks after the completion of chemotherapy, patients undergo definitive radiotherapy for about 7 weeks. After radiotherapy, patients who did not achieve complete remission after chemotherapy may undergo surgery. Patients are followed monthly for 1 year, then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, previously untreated stage IIB, III, or IV carcinoma of the nasopharynx Metastatic disease must be limited to site amenable to curative irradiation or surgical resection Locally recurrent disease after surgery allowed Evaluable disease No prior head and neck cancer, unless treated solely by surgery

PATIENT CHARACTERISTICS: Age: Any age Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3000/mm3 OR Absolute neutrophil count at least 1000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (transfusion allowed) Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT/SGPT no greater than 1.5 times ULN (no greater than 2.5 times ULN if alkaline phosphatase no greater than ULN) Alkaline phosphatase no greater than 2.5 times ULN (no greater than 4 times ULN if SGOT/SGPT no greater than ULN) Alkaline phosphatase has no ULN if known bony invasion present and all other hepatic enzymes normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: No significant cardiovascular disease Pulmonary: No significant pulmonary disease Other: No other concurrent or prior malignancy within the past 3 years except limited basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No grade 2 or worse peripheral neuropathy No other serious illness or medical condition Adequate and nutritionally balanced enteral intake No requirement for intravenous alimentation as primary source of calories Able to tolerate 3-4 liters of IV saline per day Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for nasopharyngeal cancer Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for nasopharyngeal cancer Surgery: See Disease Characteristics Recovered from prior surgery Other: Recovered from prior diagnostic or therapeutic procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Study Chair — NCI - Investigational Drug Branch
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts